CLINICAL TRIAL: NCT04403191
Title: Comparative Study Between Ondansetron, Isopropyl Alcohol Inhalation and Super Hydration in Treatment of Postoperative Emesis After Laparoscopic Appendectomy
Brief Title: Usage of Multiple Drugs in Treatment of Postoperative Vomiting After Laparoscopic Appendectomy
Status: Completed | Type: Observational
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ICU-10-20
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-03

CONDITIONS: to Treat the Vomiting Frequently Occur Post-laparoscopic by Different Anti Emetic Drugs
MeSH Terms: interventions — Ondansetron; 2-Propanol; Inhalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Group A: received ondansetron 4 mg intravenous immediately once reached to I.C.U and another same dose after 6 hours
  Interventions: Drug: Ondansetron; Procedure: laparoscopic appendectomy
- Group B: received isopropyl alcohol 70% inhalation every 15 min for 4 times then repeated after 6 hours
  Interventions: Drug: isopropyl alcohol 70% inhalation; Procedure: laparoscopic appendectomy
- Group C: received intravenous normal saline at rate of 20 ml/kg over 30 minute and repeated by the same dose after 6 hours.
  Interventions: Procedure: laparoscopic appendectomy

INTERVENTIONS:
Drug: Ondansetron — ondansetron 4 mg intravenous immediately once reached to I.C.U and another same dose after 6 hours while patients of group
  Groups: Group A
Drug: isopropyl alcohol 70% inhalation — inhalation every 15 min for 4 times then repeated after 6 hours
  Groups: Group B
Procedure: laparoscopic appendectomy — all patients received post operatively after laparoscopic appenectomy

SUMMARY:
To compare and evaluate the antiemetic effect and the safety of ondansetron, inhalational isopropyl alcohol and super hydration on adult patients after laparoscopic appendectomy.

DETAILED DESCRIPTION:
This prospective double-blind study done on 240 patients admitted to surgical I.C.U after laparoscopic appendectomy. Those who had preoperative Koivuranta vomiting score of more than 3 enrolled in our study. Every group contains 80 patients. Patients of group A received ondansetron 4 mg intravenous immediately once reached to I.C.U and another same dose after 6 hours while patients of group B received isopropyl alcohol 70% inhalation every 15 min for 4 times then repeated after 6 hours. The last group C received intravenous normal saline at rate of 20 ml/kg over 30 minute and repeated by the same dose after 6 hours. The duration of the study was 24 hours post-operatively. As PONV is self-limited within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

postoperative nausea and vomiting

Exclusion Criteria:

systemic disease as diabetes or hypertension local gastric diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 240 patients admitted to surgical I.C.U of King Abdul-Aziz specialist hospital for post-operative care after laparoscopic appendectomy surgery between March 2019 till February 2020. A Koivuranta Score to Predict Postoperative Nausea and Vomiting done preoperatively for all the patients and only those who had score of more than 3 on Koivuranta vomiting score (had more than 60% chance to develop PONV) enrolled in our study. And randomly allocated in one of three groups group A, B or C.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
numbers of vomiting attacks | for one day
  numbers of vomiting attacks recorded every 15 minutes for one day

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
To compare and evaluate the antiemetic effect and the safety of ondansetron, inhalational isopropyl alcohol and super hydration on adult patients after laparoscopic appendectomy.